CLINICAL TRIAL: NCT06341582
Title: Prediction and Evaluation by ETCOc of Neonatal Hyperbilirubinemia (PREVENT) Cohort: a Multi-center Prospective Cohort Study
Brief Title: Prediction and Evaluation by ETCOc of Neonatal Hyperbilirubinemia Cohort
Acronym: PREVENT
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Huayan Zhang, M.D., Professor, Division Chief, Guangzhou Women and Children's Medical Center
Other Study IDs: 2023-10-14
Record Dates: First submitted 2023-12-24; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Jaundice; Neonatal Hyperbilirubinemia; Hemolysis Neonatal
Keywords: Neonatal Hyperbilirubinemia; Hemolysis Neonatal; End-tidal carbon monoxide-corrected (ETCOc)
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Neonates with hemolytic hyperbilirubinemia: Neonates who are diagnosed as neonatal hyperbilirubinemia and hemolytic diseases of newborns.
  Neonatal hyperbilirubinemia is defined as the total serum bilirubin (TSB) reaching or exceeding the thresholds in aligned with the 2004 American Academy of Pediatrics (AAP) guidelines.
  Hemolytic diseases of newborns is defined as a diagnosis of ABO hemolytic diseases of newborns and/or glucose-6-phosphate dehydrogenase (G6PD) deficiency.
  Interventions: Diagnostic Test: End-tidal carbon monoxide-corrected (ETCOc)
- Neonates without hemolytic hyperbilirubinemia: Neonates who have no neonatal hyperbilirubinemia.
  Interventions: Diagnostic Test: End-tidal carbon monoxide-corrected (ETCOc)

INTERVENTIONS:
Diagnostic Test: End-tidal carbon monoxide-corrected (ETCOc) — Early postnatal ETCOc levels

SUMMARY:
The hemolytic disease of newborns (HDN) is one of the most significant risk factors for hyperbilirubinemia. Studies have shown that end-tidal carbon monoxide-corrected (ETCOc) correlated with the rate of bilirubin production in the body and thus can be a good surrogate to quantify hemolysis and identifying the high-risk infants. However, there is insufficient clinical evidence regarding the early prediction of hemolytic hyperbilirubinemia using ETCOc. This study hypothesizes that early postnatal ETCOc levels are significantly associated with the risk of hemolytic hyperbilirubinemia requiring treatments within 14 days after birth, and early postnatal ETCOc can be a good indicator for early prediction of hemolysis. In addition, the investigators aim to investigate the relationship between the characteristics of treatments for hyperbilirubinemia and ETCOc.

DETAILED DESCRIPTION:
Study design: this study is a multi-center, prospective observational cohort study on neonatal jaundice. Eligible participants will be enrolled in the well-baby nursery and neonatal intensive care units (NICU). Transcutaneous bilirubin and/or total serum bilirubin (TCB/TSB) will be measured as per clinical practice and simultaneous ETCOc (within time intervals ≤3 hours) will be monitored until (1) the newborn is discharged with the mother, or (2) until 72 hours after birth or (3) requiring the treatments for hyperbilirubinemia (phototherapy and/or exchange transfusion) (whichever comes first). For infants who do not require treatments for hyperbilirubinemia (phototherapy and/or exchange transfusion) during the stay in well-baby nursery or in the NICU within 72 hours after birth, they will be followed up via telephone or outpatient clinic visits during the first 14 days of life (DOL).

The primary outcome is the first occurrence of hemolytic hyperbilirubinemia requiring treatments within DOL14. For participants who have the primary outcome occurred within DOL14, follow-up calls/visits will continue until DOL28 to record the readmissions due to hyperbilirubinemia within 28 DOL . The secondary outcomes are 1) the incidence of hemolytic diseases of newborns; 2) characteristics of treatment for hemolytic hyperbilirubinemia: postnatal age when requiring the treatment, levels of TCB/TSB/ETCOc during hospitalization, length of stay, length of phototherapy, courses of phototherapy, exchange of transfusion, the use of intravenous immunoglobulin; 3) characteristics of readmission for hyperbilirubinemia in 28 DOL: readmission for hyperbilirubinemia in 28 DOL, postnatal age when readmitted, TCB/TSB levels when readmitted

Exposures and measurements:

1. Early postnatal (≤72 hours) ETCOc levels
2. ETCOc levels within 14 days after birth
3. ETCOc levels before each phototherapy and/or exchange transfusion treatment
4. ETCOc levels when stopping phototherapy and/or exchange transfusion treatment

Covariates and characteristics: covariates will be collected including maternal and prenatal history (e.g., mother's blood type [ABO and Rh type], G6PD deficiency status, etc.), family history (e.g., history of hemolytic diseases in the previous newborn, history of NHB treatment in the previous newborn, etc.). Clinical characteristics include demographic characteristics (e.g., gestational age, birth weight), infant's blood type (ABO and Rh type), the status of G6PD deficiency,ABO incompatibility and hemolysis, feeding history and other risk factors (e.g., early discharge after birth, excessive weight loss and the presence of hematoma) as well as data related to the primary and secondary outcomes.

For analysis, this study will examine the association between early postnatal ETCOc and the incidence of hemolytic hyperbilirubinemia, and the relation of ETCOc levels with the characteristics of treatments for hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

* Infants who are born at gestational age ≥35 weeks and with a birth weight ≥2000 grams within 72 hours after birth
* Infants who are born at study centers
* Infants with the informed consent obtained from the parents or legal guardians

Exclusion Criteria:

* Immediate requirement of respiratory support after birth (e.g., mechanical ventilation, nasal high-flow cannula oxygen therapy)
* Mothers who have active tobacco smoking or continuous environmental tobacco exposure during pregnancy
* Major congenital anomalies (e.g., cardiac or lung abnormalities, lethal chromosomal defects)
* The presence of injury of nasal mucosa, choanal atresia or Pierre Robin Sequence

Ages: 1 Hour to 72 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The eligible study population will be screened in the well-baby nursery or the neonatal intensive care unit (NICU).
Sampling Method: Probability Sample
Enrollment: 2700 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of hemolytic hyperbilirubinemia within 14 days of life (DOL) | Within 14 days of life (DOL)
  The incidence of neonatal hyperbilirubinemia and hemolytic diseases of newborns

SECONDARY OUTCOMES:
The incidence of neonatal hyperbilirubinemia within 14 days of life (DOL) | Within 14 days of life (DOL)
  The diagnosis of neonatal hyperbilirubinemia as per the 2004 AAP guidelines
The incidence of hemolytic diseases of newborns within 14 days of life (DOL) | Within 14 days of life (DOL)
  The diagnosis of ABO hemolytic diseases of newborns and/or G6PD deficiency

OTHER OUTCOMES:
The rate of readmission due to neonatal hyperbilirubinemia within 28 days of life (DOL) | Within 28 days of life (DOL)
  The readmission rate due to neonatal hyperbilirubinemia for neonates who are previously admitted because of neonatal hyperbilirubinemia within 28 DOL

CONTACTS AND LOCATIONS:
Overall Officials: Huayan Zhang, M.D., Principal Investigator — Guangzhou Women and Children's Medical Center
Locations (7):
- China (7):
  - Dongguan Maternity and Child Healthcare Hospital, Dongguan, Guangdong
  - Foshan Shunde Women and Children Health Care Hospital, Foshan, Guangdong
  - Guangdong Maternity and Child Healthcare Hospital, Guangzhou, Guangdong
  - The First affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The First Affiliated Hospital of Jinan University, Guangzhou Overseas Chinese Hospital, Guangzhou, Guangdong
  - Shenzhen Maternity and Child Healthcare Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.